CLINICAL TRIAL: NCT01217554
Title: Kinematical Evaluation of Lumbar Rotation in Neutral Position and Full Flexion in Sitting and Standing in Patients With Non-specific Chronic Low Back Pain
Brief Title: Kinematical Evaluation of Lumbar Rotation in Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Uzi Milman, Director, Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL., Clalit Health Services
Other Study IDs: K09158ctil
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Disability; Kinematic measures
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- age-matched healthy male participants: age-matched healthy male participants without LBP
- participants with non specific chronic LBP: male participants with non specific chronic LBP

SUMMARY:
Low back pain (LBP) is considered one of the most common musculoskeletal disorders in modern society, resulting in substantial costs to society. Factors associated with the development of low back pain include poor posture, strenuous work with the body, inadequate non ergonomic work and traumas.

Rotation movement pattern of the lumbar spine in different positions is essential aspect in understanding the LBP Pathophysiology. Rotation coupled with forward bending (flexion) is a dominant factor which could increase the risk LBP and disc prolapse. There is also a decline in range of motion (ROM) of rotation in forward bending (flexion) compared to neutral position during sitting and standing.

In addition,lumbar rotation movement patterns differ in population with LBP compared to asymptomatic individuals. Healthy individuals exhibit rotation accompanied by consistent coupled movement patterns of lateral bending in the opposite direction at thr upper levels, and by lateral bending in tge same direction at the lower levels . while Chronic LBP patients exhibit non consistent patterns altered from those of the normal population.

DETAILED DESCRIPTION:
According to the investigators, Kinematic measures of velocity and acceleration of lumbar rotation in neutral position and full flexion in sitting and standing did not studied yet. Evaluating these parameters, in addition to ROM and plains evaluation in the LBP population, compared to healthy population will contribute a lot in understanding this issue.

ELIGIBILITY:
Inclusion Criteria:

* non specific chronic LBP (three months or more)
* Insured by Clalit Health Care Services
* Signed informed consent

Exclusion Criteria:

* History of spinal /pelvic surgery.
* Trauma or fracture of spine /pelvis.
* Inflammatory diseases of spine.
* radiation to lower extremities .
* Neurological disease.
* malignancy disease. structural deformity of vertebral structures(scoliosis, kyphosis).

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals referred to physiotherapy for LBP
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Kinematic measures of rotation movement of the lumbar spine | one evaluation at enrollement
  Kinematic measures of rotation movement of the lumbar spine (plain, range, angular velocity and acceleration) will be measured by using Lumbar motion monitor Industrial (ILMM) .
Disability Questionnaire | one evaluation at enrollement
  Roland Morris Disability Questionnaire
pain assessment | one evaluation at enrollement
  Visual analog scale for pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Noga Maor Rougin, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL; ALAA HAJ, BA, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL; Uzi Milman, MD, Study Director — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL
Locations (1):
- Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel